CLINICAL TRIAL: NCT02282072
Title: PINS Stimulator System for Deep Brain Stimulation of the Nucleus Accumbens to Treat Severe Opioid Addiction
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Pins Medical Co., Ltd (Industry)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PINS-003
Record Dates: First submitted 2014-09-26; First posted 2014-11-04 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-08

CONDITIONS: Opioid Addiction
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deep Brain Stimulation (Active Comparator): Stimulator is ON
  Interventions: Device: Deep brain stimulation：PINS Stimulation System
- Placebo (Sham Comparator): Stimulator is OFF
  Interventions: Device: Deep brain stimulation：PINS Stimulation System

INTERVENTIONS:
Device: Deep brain stimulation：PINS Stimulation System
  Other Names: Non-rechargeable Implanted device

SUMMARY:
The purpose of this study is to verify efficacy and safety of a bilateral deep brain stimulation (DBS) of the Nucleus accumbens (NAc) as a treatment option for severe opioid addiction.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old.
2. In accordance with the diagnostic standards of DSM-IV & ICD-10 for addicted and DSM-IV for abstinence.
3. Qualitative urine detection for opioids showing positive result.
4. Cleared for 8 to 36 hours after their last drug taking.
5. Fully understood and signed on informed consent.

Exclusion Criteria:

1. Person with consciousness disorder on opioid abstinence, seriously aggressive, heavily dehydrated and intending to commit suicide.
2. Patients with serious liver and kidney dysfunction, pulmonary decompensation, or complicated with serious damage in other systems.
3. Patients with serious infectious disease.
4. Patients with history of serious neurological or psychiatrical diseases.
5. Person with history of HIV infection or serious malnutrition.
6. Dependent upon and addicted to multiple drugs.
7. Attended some other drug trials within one month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Schedule for the Assessment of Negative Symptoms (SANS) | 6 month

SECONDARY OUTCOMES:
Chronic Hunger Scale | 6 month
Beck Depression Inventory | 6 month
Buss & Perry Aggression Questionnaire | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Li Luming, PhD, Study Chair — Tsinghua University
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China